CLINICAL TRIAL: NCT06778694
Title: Comparative Effects of Motor Control and Isolated Strengthening Lumbar Exercises on Functional Outcomes in Patients with Chronic Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Faisalabad (Other)
Responsible Party: Principal Investigator, Hafiza Ayesha Aslam, Hafiza Ayesha Aslam, University of Faisalabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILEX MCE
Record Dates: First submitted 2025-01-12; First posted 2025-01-16 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Chronic Low-back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Motor control exercises
  Interventions: Other: Motor control exercises
- Group 2 (Experimental): Isolated strengthening lumbar exercises
  Interventions: Other: Isolated strengthening lumbar exercises

INTERVENTIONS:
Other: Motor control exercises — Bridging Dead bug Plank Pelvic tilts Squatting and lunges
  Arms: Group 1
Other: Isolated strengthening lumbar exercises — Child pose Mckenzie Lat pull down Russian twist
  Arms: Group 2

SUMMARY:
Comparative effects of motor control and isolated strengthening lumbar exercises on functional outcomes in patients with chronic low back pain

DETAILED DESCRIPTION:
As there is an increasing population of low back pain because of the stress and workload that lead to poor posture. Poor posture leads to tightening of flexor muscles and weakness of lumbar extensors that knowns as lower cross syndrome and it will become the chronic low back pain if not treated on time. Most of the therapist only work on the pain management but not focus on the functional outcome of the patient so the isolated lumbar extensor strengthening exercises and motor control exercises should be evaluated to know the effectiveness in improving the functional outcome of patients.

To compare the effects of motor control and isolated strengthening lumbar exercises on functional outcome in patients with chronic low back pain. A randomized controlled trial with a sample of 35 patients with chronic low back pain will be taken from Physiotherapy OPDs of Madinah Teaching Hospital, Allied hospital, In motion physiotherapy clinic and The Physio Rehab clinic. Participants will be randomly divided into two groups using convenient sampling technique. Both groups will be experimental groups. Patients in Group A will do Motor control exercises. Patients in Group B will do isolated strengthening lumbar exercises. Hot pack will be applied for 15 minutes and Ultrasound therapy (1MHz) for 3-5 minutes as baseline treatment in both groups. Patients will be included based on inclusion and exclusion criteria. Assessment will be done by using NPRS and Oswestry disability Index Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* LBP for more than 3 months

Both male and females.

Age between 20-50 years old.

Moderate to severe pain (VAS; 3-7)

Currently seeking care for LBP.

Exclusion Criteria:

* Spinal surgery

Pregnancy

Prostatectomy

Engaged in any sports activities

Any evidence of nerve root compression

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
NPRS | Baseline and after 2 and 4 weeks of treatment
  Comparison on effect of pain

SECONDARY OUTCOMES:
Oswestry disability Questionnaire | Baseline and after 2 and 4 weeks of treatment
  Comparison on functional outcome

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saragiotto BT, Maher CG, Yamato TP, Costa LO, Menezes Costa LC, Ostelo RW, Macedo LG. Motor control exercise for chronic non-specific low-back pain. Cochrane Database Syst Rev. 2016 Jan 8;2016(1):CD012004. doi: 10.1002/14651858.CD012004. PMID 26742533
- [Background] Fanuscu A, Oz M, Ozel Asliyuce Y, Turhan E, Ulger O. Effects of Clinic-based and Telerehabilitation-based Motor Control Exercises in Individuals with Chronic Low-back Pain: A Randomized Controlled Trial With 3-Month Follow-up. Clin J Pain. 2024 Dec 1;40(12):700-708. doi: 10.1097/AJP.0000000000001245. PMID 39285790
- [Background] Steele J, Bruce-Low S, Smith D, Jessop D, Osborne N. Isolated Lumbar Extension Resistance Training Improves Strength, Pain, and Disability, but Not Spinal Height or Shrinkage ("Creep") in Participants with Chronic Low Back Pain. Cartilage. 2020 Apr;11(2):160-168. doi: 10.1177/1947603517695614. Epub 2017 Feb 1. PMID 29156985
- [Background] Steele J, Fisher J, Bruce-Low S, Smith D, Osborne N, Newell D. Variability in Strength, Pain, and Disability Changes in Response to an Isolated Lumbar Extension Resistance Training Intervention in Participants with Chronic Low Back Pain. Healthcare (Basel). 2017 Oct 16;5(4):75. doi: 10.3390/healthcare5040075. PMID 29035297
- [Background] Fortin M, Rye M, Roussac A, Montpetit C, Burdick J, Naghdi N, Rosenstein B, Bertrand C, Macedo LG, Elliott JM, Dover G, DeMont R, Weber MH, Pepin V. The Effects of Combined Motor Control and Isolated Extensor Strengthening versus General Exercise on Paraspinal Muscle Morphology, Composition, and Function in Patients with Chronic Low Back Pain: A Randomized Controlled Trial. J Clin Med. 2023 Sep 12;12(18):5920. doi: 10.3390/jcm12185920. PMID 37762861